CLINICAL TRIAL: NCT02082977
Title: A Phase I Open-label, Dose Escalation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Activity of GSK2816126 in Subjects With Relapsed/Refractory Diffuse Large B Cell Lymphoma, Transformed Follicular Lymphoma, Other Non-Hodgkin's Lymphomas, Solid Tumors and Multiple Myeloma
Brief Title: A Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Activity of GSK2816126 in Subjects With Relapsed/Refractory Diffuse Large B Cell Lymphoma, Transformed Follicular Lymphoma, Other Non-Hodgkin's Lymphomas, Solid Tumors and Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The maximal dose and schedule attained with GSK2816126 has shown insufficient evidence of clinical activity, and does not justify further clinical investigation
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 117208; 2013-001585-42 (EudraCT Number)
Record Dates: First submitted 2014-01-16; First posted 2014-03-11 (Estimated); Results first posted 2019-06-28 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Cancer; Neoplasms
Keywords: Refractory; Phase I study, dose escalation study; diffuse large B cell lymphoma; Relapsed; Solid tumors; transformed follicular lymphoma; Multiple myeloma; GSK2816126; Non-Hodgkin's lymphoma
MeSH Terms: conditions — Neoplasms; Lymphoma, Large B-Cell, Diffuse; Recurrence; Multiple Myeloma; Lymphoma, Non-Hodgkin | interventions — GSK-2816126

STUDY DESIGN:
Intervention Model Description: Subjects will receive escalating doses of GSK2816126 in Part 1 of the study. Subjects enrolled in Part 2 will receive recommended Phase II dose (RP2D) based on Part 1 of the study.
Masking Description: This will be an open-label study. Hence, there will be no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Part 1:GSK2816126 50 mg twice-weekly (Experimental): Eligible subjects will receive GSK2816126 with a starting dose of 50 milligrams (mg) twice-weekly, as an intravenous solution for 28 days (3 weeks on/1 week off).
  Interventions: Drug: GSK2816126
- Part 1:GSK2816126 100 mg twice-weekly (Experimental): Eligible subjects will receive GSK2816126 with a dose of 100 mg twice-weekly, as an intravenous solution for 28 days (3 weeks on/1 week off).
  Interventions: Drug: GSK2816126
- Part 1:GSK2816126 200 mg twice-weekly (Experimental): Eligible subjects will receive GSK2816126 with a dose of 200 mg twice-weekly, as an intravenous solution for 28 days (3 weeks on/1 week off).
  Interventions: Drug: GSK2816126
- Part 1:GSK2816126 400 mg twice-weekly (Experimental): Eligible subjects will receive GSK2816126 with a dose of 400 mg twice-weekly, as an intravenous solution for 28 days (3 weeks on/1 week off).
  Interventions: Drug: GSK2816126
- Part 1:GSK2816126 800 mg twice-weekly (Experimental): Eligible subjects will receive GSK2816126 with a dose of 800 mg twice-weekly, as an intravenous solution for 28 days (3 weeks on/1 week off).
  Interventions: Drug: GSK2816126
- Part 1:GSK2816126 1200 mg twice-weekly (Experimental): Eligible subjects will receive GSK2816126 with a dose of 1200 mg twice-weekly, as an intravenous solution for 28 days (3 weeks on/1 week off).
  Interventions: Drug: GSK2816126
- Part 1:GSK2816126 1800 mg twice-weekly (Experimental): Eligible subjects will receive GSK2816126 with a dose of 1800 mg twice-weekly, as an intravenous solution for 28 days (3 weeks on/1 week off).
  Interventions: Drug: GSK2816126
- Part 1:GSK2816126 2400 mg twice-weekly (Experimental): Eligible subjects will receive GSK2816126 with a dose of 2400 mg twice-weekly, as an intravenous solution for 28 days (3 weeks on/1 week off).
  Interventions: Drug: GSK2816126
- Part 1:GSK2816126 3000 mg twice-weekly (Experimental): Eligible subjects will receive GSK2816126 with a dose of 3000 mg twice-weekly, as an intravenous solution for 28 days (3 weeks on/1 week off).
  Interventions: Drug: GSK2816126
- Part 2: All subjects (Experimental): Subjects with Germinal Center B-cell-like Diffuse Large B-cell Lymphoma (GCB-DLBCL)-mutant and wild type, Transformed Follicular Lymphoma (TFL)-mutant and wild type as well as with multiple myeloma (MM) will be enrolled in Part 2 of the study. Subjects enrolled in Part 2 will receive recommended Phase II dose (RP2D).
  Interventions: Drug: GSK2816126

INTERVENTIONS:
Drug: GSK2816126 — GSK2816126 will be supplied as a solution containing 15 milligram per milliliter (mg/mL) GSK2816126 in water for injection.

SUMMARY:
This is an open-label, multicenter, 2-part study to determine the recommended Phase 2 dose (RP2D) for GSK2816126 given twice weekly by intravenous (IV) infusion. Part 1 will be conducted in adult subjects with relapsed/refractory diffuse large B cell lymphoma (DLBCL), transformed follicular lymphoma (tFL), other Non-Hodgkin's lymphomas (NHL), solid tumors (including castrate resistant prostate cancer) and multiple myeloma (MM) to determine the safety and tolerability of GSK2816126. Expansion cohorts (Part 2) are planned to further explore clinical activity of GSK2816126 at the RP2D in subjects with Enhancer of Zeste 2 (EZH2) wild type and EZH2 mutant positive germinal center B-cell like diffuse large B cell lymphoma (GCB-DLBCL), tFL and MM.

ELIGIBILITY:
Part 1 Inclusion Criteria

* Provided signed written informed consent
* Males and females >=18 years of age (at the time consent is obtained).
* Tumor type criteria: relapsed/refractory non-Hodgkin's lymphoma (NHL) that meets one of the following criteria:
* Germinal Center B cell Diffuse large B cell lymphoma (GCB-DLBCL) relapsed or refractory to at least one prior regimen (e.g., rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone [R-CHOP]) AND not a candidate for standard salvage regimens or autologous or allogeneic stem cell transplant. Local confirmation of lymphoma subtype (e.g. GCB-DLBCL) is allowed for enrollment but must be confirmed through central laboratory testing.
* Solid tumors that meet the following criteria: Measurable disease by Response Evaluation Criteria In Solid Tumors 1.1 (RECIST) in at least 1 site. For Castrate Resistant Prostate Cancer (CRPC) measurable disease can also include Prostate Specific Antigen (PSA) level. Disease progression with the last line of therapy and at least one prior standard of care regimens, or tumor for which there is no approved therapy, or for which standard therapy is unsuitable or refused. Mutation Status: Solid tumor types, other than prostate, must have a one of the following EZH2 inhibitor sensitizing mutations as determined via local testing: An activating mutation in EZH2 (Y641F/C/S/H/N, A677V/G, and/or A687V; Loss of a component of the SWI/SNF complex, including, but not limited to, ARID1A, SMARCB1 (aka SNF5/INI1/BAF47), SMARCA4 (aka BRG1), or PBRM1 (aka PB1) as determined by molecular testing (bi-allelic loss or mutation) or immunohistochemistry; Loss of BAP1 (ubiquitin carboxy-terminal hydrolase) as determined by molecular testing (bi-allelic loss or mutation) or immunohistochemistry
* CRPC subjects: Must have measurable disease by either: RECIST1.1 or a minimum PSA of 5 nanogram/milliliter; Disease progression on last line of therapy and must have progressed on abiraterone, enzalutamide, or taxane chemotherapy; Subjects may continue GnRH agonists; Small cell prostate cancer is eligible
* For all subjects: Availability of archival tissue, or willingness to undergo fresh biopsy if archival tissue is not available.
* Must have a pre-existing central venous access such as a port, Hickmann catheter or a peripherally inserted central catheter (PICC line) or be willing and able to have one inserted.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Men with a female partner of childbearing potential must have either had a prior bilateral vasectomy with resultant azoospermia, bilateral orchiectomy, or must agree to use one of the contraception methods listed in protocol from the time of the first dose of study medication until at least 2 weeks (14 days) after the last dose of study treatment due to the long elimination phase of study drug.
* A female subject is eligible to participate ifs she is of: Non-child bearing potential as described in the protocol; OR Child bearing potential and agrees to use effective contraception as described in the protocol, for an appropriate period of time (as determined by the product label) prior to the start of dosing to sufficiently minimize the risk of pregnancy and for at least 2 weeks (14 days) following the last dose of study treatment. Women of childbearing potential must have a negative serum pregnancy test within 7 days of first dose of study treatment followed by negative urine or serum pregnancy test once every 4 weeks (prior to next dose cycle) thereafter.- Adequate organ system function as defined in the protocol.

Part 2 Inclusion Criteria

* In addition to inclusion criteria listed for Part 1, Part 2 will enroll GCB-DLBCL tFL and MM subjects only. Relapsed and/or refractory MM or tFL that have failed prior standard therapy and for which there is no standard salvage regimen
* Lymphoma subjects will be required to undergo EZH2 mutation testing. This will require availability of archival tissue, or willingness to undergo fresh biopsy, for central testing of EZH2 mutation status.
* Based on the results of the mutation test, lymphoma subjects may be enrolled in one of four cohorts: GCB-DLBCL EZH2 mutant cohort: Tumors must contain one, or more, of the following EZH2 activating mutations: Y641F; Y641N; Y641S; Y641H; Y641C; A677G; and/or A687V. GCB-DLBCL EZH2 wild type cohort: Tumors that do not contain one of the above mutations; Subjects with tumors harboring EZH2 mutations other than the seven outlined above will be enrolled in the EZH2 wild type cohort. tFL EZH2 mutant cohort: Tumors must contain one, or more, of the following EZH2 activating mutations: Y641F; Y641N; Y641S; Y641H; Y641C; A677G; and/or A687V. tFL EZH2 wild type cohort: Tumors that do not contain one of the above mutations; Subjects with tumors harboring EZH2 mutations other than the seven outlined above will be enrolled in the EZH2 wild type cohort

Part 1 and 2 Exclusion Criteria

* Receiving any cancer therapy within 2 weeks of first dose (including surgery, and/or tumor embolization) Note: the following are allowed: Corticosteroids to control systemic or local symptoms, up to a dose of 10 mg prednisone or equivalent daily and stable for at least 7 days prior to enrollment. Subjects with prostate cancer may remain on GnRH agonists. Other hormonal therapies (e.g., bicalutamide, abiraterone and enzlutimide) for prostate cancer must be stopped 4 weeks prior to enrolment.

Note: the following are NOT allowed: Chemotherapy regimens with delayed toxicity within the last 3 weeks. Nitrogen mustards, Melphalan, Monoclonal antibody or Nitrosourea within the last 6 weeks.

* Received an investigational anti-cancer drug within 6weeks, or within 5 half-lives (whichever is shorter) of the first dose of study drug(s). A minimum of 14 days must have passed between the last dose of prior investigational agent and the first dose of study drug.
* Current use of a prohibited medication per protocol or expected to require any of these medications during treatment with study drug.
* Known Human Immunodeficiency Virus, or serological evidence for Hepatitis B (positive hepatitis B surface antigen [HBsAg]), or chronic Hepatitis C infection. For subjects who are negative for HBsAg, but Hepatitis B core Antibody [HBcAB] positive, a HBV DNA (viral load) test will be performed and if negative are eligible. Subjects with positive Hepatitis C antibody serology with a negative HCV ribonucleic acid (RNA) test results are eligible.
* Concurrent use of therapeutic warfarin is allowed. However, anticoagulants that do not have reversal agents available are prohibited.
* Any major surgery, radiotherapy or immunotherapy within the 4 weeks prior to first dose of study drug, or palliative radiotherapy to a single symptomatic lesion within the 2 weeks prior to first dose of study drugs.
* Subjects with prior allogeneic transplant are excluded: however, subjects who have previously received an autologous stem cell transplant are allowed if a minimum of 100 days has elapsed from the time of transplant and the subject has recovered from transplant-associated toxicities prior to the first dose of GSK2816126
* Unresolved toxicity greater than Grade 1 National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4 from previous anti-cancer therapy, with the exception of alopecia and peripheral neuropathy. Lymphoma subjects with <= Grade 3 lymphopenia can be enrolled at the discretion of the investigator.
* Packed red blood cell or platelet transfusion within 7 days of screening laboratory tests.
* Psychological, familial, sociological or geographical conditions that do not permit compliance with the protocol.
* Cardiac exclusion criteria: History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within the past 6 months prior to first dose of study drug; QTcF> 450 milliseconds (msec); Uncontrolled arrhythmias. Subjects with rate controlled atrial fibrillation for >1 month prior to first dose of study drug may be eligible; Class II, III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drug or their excipients.
* Pregnant or lactating female.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Uncontrolled diabetes or other medical condition that may interfere with assessment of toxicity.
* Central nervous system (CNS) metastases, with the following exception: Subjects who have previously treated CNS metastases, are asymptomatic, and have no requirement for steroids at least 14 days prior to first dose of study drug; Subjects with carcinomatous meningitis are excluded regardless of clinical stability.
* Invasive malignancy or history of invasive malignancy other than disease under study: any other invasive malignancy from which the subject has been disease-free for more than 2 years and, in the opinion of the principal investigator and GSK Medical Monitor, will not affect the evaluation of the effects of this clinical trial treatment on currently targeted malignancy, can be included in this clinical trial; Curatively treated non-melanoma skin cancer and any carcinoma-in-situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-04-24 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (2):
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, New York, New York
- GSK Investigational Site, Villejuif, France
- United Kingdom (2):
  - GSK Investigational Site, Sutton, Surrey
  - GSK Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20101

REFERENCES:
- [Background] Yap TA, Winter JN, Giulino-Roth L, Longley J, Lopez J, Michot JM, Leonard JP, Ribrag V, McCabe MT, Creasy CL, Stern M, Pene Dumitrescu T, Wang X, Frey S, Carver J, Horner T, Oh C, Khaled A, Dhar A, Johnson PWM. Phase I Study of the Novel Enhancer of Zeste Homolog 2 (EZH2) Inhibitor GSK2816126 in Patients with Advanced Hematologic and Solid Tumors. Clin Cancer Res. 2019 Dec 15;25(24):7331-7339. doi: 10.1158/1078-0432.CCR-18-4121. Epub 2019 Aug 30. PMID 31471312

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2-part study in participants with relapsed/refractory diffuse large B cell lymphoma, transformed follicular lymphoma, other Non-Hodgkin's lymphomas, solid tumors and multiple myeloma (MM). In Part 1 dose escalation, participants received 50 to 3000 milligrams (mg) of GSK2816126, and Part 2 was dose expansion.
Pre-assignment Details: This study was terminated prior to the completion of Part 1 due to an unfavorable benefit risk profile. Part 2 was not conducted. Approximately 42 participants screened, of which 41 were treated in Part 1 including 20 participants with lymphoma and 21 with solid tumors, of these 22 completed, 5 died and 14 participants were withdrawn.
Groups:
- Part 1:GSK2816126 50 mg Twice-weekly: Eligible participants received GSK2816126 with a starting dose of 50 mg twice-weekly, as an intravenous solution for 28 days (3 weeks on/1 week off).
- Part 1:GSK2816126 100 mg Twice-weekly: Eligible participants received GSK2816126 with a dose of 100 mg twice-weekly, as an intravenous solution for 28 days (3 weeks on/1 week off).
- Part 1:GSK2816126 200 mg Twice-weekly: Eligible participants received GSK2816126 with a dose of 200 mg twice-weekly, as an intravenous solution for 28 days (3 weeks on/1 week off).
- Part 1:GSK2816126 400 mg Twice-weekly: Eligible participants received GSK2816126 with a dose of 400 mg twice-weekly, as an intravenous solution for 28 days (3 weeks on/1 week off).
- Part 1:GSK2816126 800 mg Twice-weekly: Eligible participants received GSK2816126 with a dose of 800 mg twice-weekly, as an intravenous solution for 28 days (3 weeks on/1 week off).
- Part 1:GSK2816126 1200 mg Twice-weekly: Eligible participants received GSK2816126 with a dose of 1200 mg twice-weekly, as an intravenous solution for 28 days (3 weeks on/1 week off).
- Part 1:GSK2816126 1800 mg Twice-weekly: Eligible participants received GSK2816126 with a dose of 1800 mg twice-weekly, as an intravenous solution for 28 days (3 weeks on/1 week off).
- Part 1:GSK2816126 2400 mg Twice-weekly: Eligible participants received GSK2816126 with a dose of 2400 mg twice-weekly, as an intravenous solution for 28 days (3 weeks on/1 week off).
- Part 1:GSK2816126 3000 mg Twice-weekly: Eligible participants received GSK2816126 with a dose of 3000 mg twice-weekly, as an intravenous solution for 28 days (3 weeks on/1 week off).
- Part 2: All Participants: Participants with Germinal Center B-cell-like Diffuse Large B-cell Lymphoma (GCB-DLBCL)-mutant and wild type, Transformed Follicular Lymphoma (TFL)-mutant and wild type as well as with MM were planned to be enrolled in Part 2 of the study. Participants enrolled in Part 2 were planned to receive recommended Phase II dose (RP2D).
Period: Part 1 (Up to 3.2 Years)
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly | Part 2: All Participants
Started | 2 | 1 | 1 | 1 | 3 | 4 | 10 | 12 | 7 | 0
Completed | 1 | 1 | 1 | 1 | 2 | 1 | 4 | 7 | 4 | 0
Not Completed | 1 | 0 | 0 | 0 | 1 | 3 | 6 | 5 | 3 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Not completed — Study closed/terminated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Period: Part 2 (Up to 3.2 Years)
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly | Part 2: All Participants
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data was not collected in Part 2 of the study as no participant was enrolled in Part 2.
Groups:
- Part 2: All Participants: Participants with Germinal Center B-cell-like Diffuse Large B-cell Lymphoma (GCB-DLBCL)-mutant and wild type, Transformed Follicular Lymphoma (TFL)-mutant and wild type as well as with MM were planned to be enrolled in Part 2 of the study. Participants enrolled in Part 2 were planned to receive recommended Phase II dose (RP2D) .
- Total: Total of all reporting groups
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly | Part 2: All Participants | Total
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 3 | 4 | 10 | 12 | 7 | 0 | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.0 (12.73) | 54.0 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant. | 56.0 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant. | 69.0 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant. | 53.3 (4.04) | 49.5 (17.18) | 61.1 (14.10) | 61.9 (14.65) | 58.4 (14.30) |  | 58.2 (13.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 7 | 4 |  | 16
  Male | 2 | 1 | 1 | 1 | 1 | 3 | 8 | 5 | 3 |  | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 |  | 1
  Asian-Central/South Asian Heritage | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 |  | 1
  White - White/Caucasian/European Heritage | 2 | 1 | 1 | 1 | 3 | 4 | 8 | 12 | 5 |  | 37
  Mixed white race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 |  | 1
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Serious Adverse Events (SAEs) and Non-serious Adverse Events (Non-SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/ incapacity, is a congenital anomaly/ birth defect, other situations and is associated with liver injury or impaired liver function. The analysis was performed on All Subjects Population which included all participants who received at least one dose of study treatment.
Time Frame: Up to 3.2 years
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 3 | 4 | 10 | 12 | 7
Participants
  Any Non-SAE | 2 | 1 | 1 | 1 | 3 | 4 | 10 | 12 | 7
  Any SAE | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 5 | 3

2. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicities (DLT)
Description: An event was considered a DLT if it occurred within first 4 weeks (28 days) of treatment, and met the criteria's for hematologic , non-hematologic, infusion reactions and other toxicities, unless it can be clearly established that the event is unrelated to treatment.
Time Frame: Up to 4 weeks
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 3 | 4 | 10 | 12 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

3. Primary Outcome: Part 1: Number of Participants Withdrawn Due to AEs
Description: A participant was considered to have completed the study if they have completed their end of study visit or if the participant died or was still in follow-up at the time the study was closed or terminated. Participants were monitored from start of the study till the development of toxicity. The data for number of participants withdrawn due to AEs have been presented.
Time Frame: Up to 3.2 years
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 3 | 4 | 10 | 12 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part 1: Number of Participants With Dose Interruptions
Description: The number of participants who had any dose interruptions have been presented.
Time Frame: Up to 3.2 years
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 3 | 4 | 10 | 12 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 5

5. Primary Outcome: Part 1: Number of Participants With Dose Reductions
Description: The number of participants who had any dose reductions have been presented.
Time Frame: Up to 3.2 years
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 3 | 4 | 10 | 12 | 7
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

6. Primary Outcome: Part 1: Number of Participants With Worst Case Change From Baseline in Clinical Chemistry Parameters
Description: Blood samples were collected for evaluation of clinical chemistry parameters including direct bilirubin, chloride, lactate dehydrogenase (LDH), total protein, urea/blood urea nitrogen (BUN) and uric acid. Baseline value was defined as the most recent, non-missing value from a local laboratory prior to the first dose of study treatment. Change from Baseline was defined as any visit value minus Baseline value. The summaries of worst case change from Baseline with respect to normal range have been presented for only those laboratory tests that are not gradable by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The number of participants with decreases to low, changes to normal or no changes from Baseline, and increases to high values have been presented. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 3.2 years
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 3 | 4 | 10 | 12 | 7
Participants
  Direct Bilirubin; To Low; n=1,1,1,1,3,4,8,12,7: number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 4 | 8 | 12 | 7
  Direct Bilirubin; To Low; n=1,1,1,1,3,4,8,12,7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin; To Normal; n=1,1,1,1,3,4,8,12,7: number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 4 | 8 | 12 | 7
  Direct Bilirubin; To Normal; n=1,1,1,1,3,4,8,12,7 | 1 | 1 | 1 | 0 | 3 | 4 | 8 | 9 | 7
  Direct Bilirubin; To High; n=1,1,1,1,3,4,8,12,7: number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 4 | 8 | 12 | 7
  Direct Bilirubin; To High; n=1,1,1,1,3,4,8,12,7 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
  Chloride; To Low;n=2,1,1,1,3,4,10,12,7 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1
  Chloride; To Normal; n=2,1,1,1,3,4,10,12,7 | 1 | 1 | 1 | 1 | 3 | 4 | 6 | 8 | 6
  Chloride; To High; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
  LDH; To Low; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  LDH; To Normal; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 1 | 1 | 3 | 4 | 8 | 9 | 5
  LDH; To High; n=2,1,1,1,3,4,10,12,7 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 2
  Total Protein; To Low n=2,1,1,1,3,4,10,12,7 | 1 | 1 | 1 | 1 | 2 | 0 | 3 | 3 | 2
  Total Protein; To Normal; n=2,1,1,1,3,4,10,12,7 | 1 | 0 | 0 | 0 | 1 | 4 | 8 | 9 | 5
  Total Protein; To High; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Urea/BUN; To Low; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Urea/BUN; To Normal; n=2,1,1,1,3,4,10,12,7 | 2 | 0 | 1 | 1 | 1 | 4 | 7 | 5 | 4
  Urea/BUN; To High; n=2,1,1,1,3,4,10,12,7 | 0 | 1 | 0 | 0 | 2 | 0 | 3 | 6 | 2
  Uric acid; To Low; n=2,1,1,1,3,4,10,12,7 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Uric acid; To Normal; n=2,1,1,1,3,4,10,12,7 | 2 | 0 | 0 | 0 | 3 | 3 | 7 | 8 | 4
  Uric acid; To High; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 4 | 2

7. Primary Outcome: Part 1: Number of Participants With Worst Case Change From Baseline in Hematology Parameters
Description: Blood samples were collected for the analysis of hematology parameters including basophils, eosinophils, hematocrit, mean corpuscular hemoglobin concentration (MCHC), mean corpuscular hemoglobin (MCH), mean corpuscular volume (MCV), monocytes, segmented (seg) neutrophils, red blood cell (RBC) count and reticulocytes. Baseline value was defined as the most recent, non-missing value from a local laboratory prior to the first dose of study treatment. Change from Baseline was defined as any visit value minus Baseline value. The summaries of worst case change from Baseline with respect to normal range have been presented for only those laboratory tests that are not gradable by CTCAE version 4.0. The number of participants with decreases to low, changes to normal or no changes from Baseline, and increases to high values have been presented. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 3.2 years
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 3 | 4 | 10 | 12 | 7
Participants
  Basophils; To Low; n=2,1,1,1,3,4,10,12,7 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 2
  Basophils; To Normal; n=2,1,1,1,3,4,10,12,7 | 1 | 1 | 1 | 1 | 2 | 3 | 9 | 9 | 5
  Basophils; To High; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils; To Low; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 2 | 0
  Eosinophils; To Normal; n=2,1,1,1,3,4,10,12,7 | 2 | 1 | 1 | 1 | 0 | 3 | 7 | 10 | 7
  Eosinophils; To High; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Hematocrit; To Low; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 4
  Hematocrit; To Normal; n=2,1,1,1,3,4,10,12,7 | 2 | 1 | 1 | 1 | 2 | 4 | 8 | 10 | 3
  Hematocrit; To High; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  MCHC; To Low; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 1 | 0 | 0 | 2 | 7 | 5 | 2
  MCHC; To Normal; n=2,1,1,1,3,4,10,12,7 | 2 | 1 | 0 | 1 | 2 | 2 | 2 | 7 | 5
  MCHC; To High; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
  MCH; To Low; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  MCH; To Normal; n=2,1,1,1,3,4,10,12,7 | 2 | 1 | 1 | 0 | 2 | 4 | 7 | 11 | 7
  MCH; To High; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0
  MCV; To Low; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  MCV; To Normal; n=2,1,1,1,3,4,10,12,7 | 1 | 1 | 1 | 1 | 2 | 3 | 9 | 11 | 7
  MCV; To High; n=2,1,1,1,3,4,10,12,7 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Monocytes; To Low; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
  Monocytes; To Normal; n=2,1,1,1,3,4,10,12,7 | 2 | 1 | 1 | 1 | 2 | 4 | 5 | 9 | 5
  Monocytes; To High; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 1
  Seg Neutrophils; To Low; n= 0,0,0,0,0,0,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Seg Neutrophils; To Low; n= 0,0,0,0,0,0,0,0,1 |  |  |  |  |  |  |  |  | 0
  Seg Neutrophils; To Normal; n= 0,0,0,0,0,0,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Seg Neutrophils; To Normal; n= 0,0,0,0,0,0,0,0,1 |  |  |  |  |  |  |  |  | 1
  Seg Neutrophils; To High; n= n= 0,0,0,0,0,0,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Seg Neutrophils; To High; n= n= 0,0,0,0,0,0,0,0,1 |  |  |  |  |  |  |  |  | 0
  RBC count; To Low; n=2,1,1,1,3,4,10,12,7 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 3
  RBC count; To Normal; n=2,1,1,1,3,4,10,12,7 | 1 | 1 | 1 | 1 | 3 | 4 | 6 | 8 | 4
  RBC count; To High; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Reticulocytes; ; To Low; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 0 | 1 | 1 | 1 | 5 | 2 | 3
  Reticulocytes; To Normal; n=2,1,1,1,3,4,10,12,7 | 2 | 1 | 1 | 0 | 2 | 3 | 5 | 10 | 4
  Reticulocytes; To High; n=2,1,1,1,3,4,10,12,7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

8. Primary Outcome: Part 1:Number of Participants With Abnormal Values for Vital Signs
Description: Vital sign measurements includes systolic blood pressure (SBP), diastolic blood pressure (DBP), body temperature and heart rate. Vital signs were measured after resting for at least 5 minutes in a semi-supine position. The number of participants with abnormal findings for vital signs have been presented.
Time Frame: Up to 3.2 years
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 3 | 4 | 10 | 12 | 7
Participants
  SBP | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0
  DBP | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 5 | 0
  Heart rate | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
  Body temperature | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Part 1: Number of Participants With Abnormal Findings for Electrocardiogram (ECG) Parameters
Description: Single measurements of 12-lead ECGs were obtained a semi-recumbent or semi-supine position after at least a 5 minutes rest using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT and corrected QT (QTc) intervals. The number of participants with abnormal, abnormal-not clinically significant (NCS), and abnormal-clinically significant (CS) worst case Post Baseline findings have been presented.
Time Frame: Up to 3.2 years
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 3 | 4 | 10 | 12 | 7
Participants
  Abnormal; NCS | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 6 | 2
  Abnormal; CS | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
  Abnormal | 2 | 0 | 0 | 1 | 1 | 2 | 5 | 5 | 4

10. Primary Outcome: Part 2: Percentage of Participants Achieving Overall Response Rate
Description: Overall response rate is defined as percentage of participants achieving complete response and partial response per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 3.2 years
Population: All Subjects Population. Data was not collected in Part 2 as no participant was enrolled in Part 2.
Groups:
- Part 2: All Participants: Participants with GCB-DLBCL-mutant and wild type, TFL-mutant and wild type as well as participants with MM were planned to be enrolled in Part 2 of the study. Participants enrolled in Part 2 were planned to receive RP2D .
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

11. Secondary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration (AUC [0-t]) Following Single and Repeat Dose Administration of GSK2816126
Description: Blood samples were collected from participants for pharmacokinetic analysis including AUC (0-t) following single (Day 1) and repeat dose (Day 15) administration of GSK2816126. Pharmacokinetic analysis of GSK2816126 in Part 1 was conducted by non-compartmental methods. The analysis was performed on Pharmacokinetic Population which included all participants in the All Subject population for whom a blood sample for pharmacokinetics was analyzed and at least 1 non-missing values was obtained. NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Pre-dose, 0.5, 1, 2, (12, 18 on Day 1 only), 24, and 96 hours post-dose from start of infusion; 0.5, 1, 2, 4, 6 hours from end of infusion on Cycle 1 of Day 1 and Day 15 (Each cycle was of 28 days)
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram per milliliter
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 3 | 4 | 10 | 12 | 7
Hour*microgram per milliliter
  Day 1; n=2,1,1,1,3,4,10,12,7 | 1.20 (62) | 27.20 (NA) — NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. | 27.70 (NA) — NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. | 11.80 (NA) — NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. | 24.18 (10) | 85.72 (91) | 45.93 (23) | 92.41 (26) | 93.96 (48)
  Day 15; n=1,1,1,1,3,4,9,11,4: number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 4 | 9 | 11 | 4
  Day 15; n=1,1,1,1,3,4,9,11,4 | 3.20 (NA) — NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. | 5.70 (NA) — NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. | 7.10 (NA) — NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. | 13.10 (NA) — NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. | 25.82 (30) | 53.41 (14) | 68.72 (75) | 105.29 (29) | 158.44 (35)

12. Secondary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC [0-infinity]) Following Single Dose Administration of GSK2816126
Description: Blood samples were collected from participants for pharmacokinetic analysis including AUC (0-infinity) following single (Day 1) dose administration of GSK2816126. Pharmacokinetic analysis of GSK2816126 in Part 1 was conducted by non-compartmental methods. NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. Pharmacokinetic parameter derivation for some participants did not strictly conform to the prescribed acceptance criteria and hence data was not available for those participants.
Time Frame: Pre-dose, 0.5, 1, 2, 12, 18 , 24, and 96 hours post-dose from start of infusion; 0.5, 1, 2, 4, 6 hours from end of infusion on Cycle 1 of Day 1 (Each cycle was of 28 days)
Population: Pharmacokinetic Population. Only those participants with data available at specific time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*Microgram per milliliter
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 2 | 0 | 0 | 1 | 3 | 1 | 10 | 10 | 7
Hour*Microgram per milliliter | 1.33 (82) |  |  | 13.20 (NA) — NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. | 26.41 (12) | 60.90 (NA) — NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. | 51.15 (23) | 102.48 (28) | 103.17 (48)

13. Secondary Outcome: Part 1: Area Under the Concentration-time Curve Over the Dosing Interval (AUC [0-tau]) Following Repeat Dose Administration of GSK2816126
Description: Blood samples were collected from participants for pharmacokinetic analysis including AUC (0-tau) following repeat (Day 15) dose administration of GSK2816126. Pharmacokinetic analysis of GSK2816126 in Part 1 was conducted by non-compartmental methods. NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant.
Time Frame: Pre-dose, 0.5, 1, 2, 24, and 96 hours post-dose from start of infusion; 0.5, 1, 2, 4, 6 hours from end of infusion on Cycle 1 of Day 15 (Each cycle was of 28 days)
Population: Pharmacokinetic Population. Only those participants with data available at specific time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*Microgram per milliliter
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 4 | 9 | 11 | 4
Hour*Microgram per milliliter | 2.90 (NA) — NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. | 5.70 (NA) — NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. | 7.10 (NA) — NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. | 12.30 (NA) — NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. | 26.85 (25) | 53.66 (14) | 59.70 (25) | 111.32 (25) | 157.88 (36)

14. Secondary Outcome: Part 1: Trough (Pre-dose) Concentration at the End of Dosing Interval on the Specified Days (Ctau) Following Administration of GSK2816126
Description: Blood samples were collected from participants for pharmacokinetic analysis including Ctau following specified days (Days 8 and 15) administration of GSK2816126. Pharmacokinetic analysis of GSK2816126 in Part 1 was conducted by non-compartmental methods. NA indicates data was not available as data could not be calculated due to limited number of participants at specified data point. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Pre-dose from start of infusion till end of infusion on Cycle 1 of Day 8; Pre-dose, 0.5, 1, 2, 24, and 96 hours post-dose from start of infusion; 0.5, 1, 2, 4, 6 hours from end of infusion on Cycle 1 of Day 15 (Each cycle was of 28 days)
Population: Pharmacokinetic Population. Only those participants with data available at specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 3 | 4 | 10 | 12 | 7
Microgram per milliliter
  Day 8; n=2,1,1,1,3,4,9,11,6: number analyzed (Participants) | 2 | 1 | 1 | 1 | 3 | 4 | 9 | 11 | 6
  Day 8; n=2,1,1,1,3,4,9,11,6 | NA (NA) — NA indicates data was not available due to limited number of participants to calculate the data. | NA (NA) — NA indicates data was not available due to limited number of participants to calculate the data. | NA (NA) — NA indicates data was not available due to limited number of participants to calculate the data. | NA (NA) — NA indicates data was not available due to limited number of participants to calculate the data. | 0.10 (0) | 0.14 (79) | 0.15 (38) | 0.33 (97) | 0.41 (147)
  Day 15; n=1,1,1,1,3,4,10,11,4: number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 4 | 10 | 11 | 4
  Day 15; n=1,1,1,1,3,4,10,11,4 | NA (NA) — NA indicates data was not available due to limited number of participants to calculate the data. | NA (NA) — NA indicates data was not available due to limited number of participants to calculate the data. | NA (NA) — NA indicates data was not available due to limited number of participants to calculate the data. | NA (NA) — NA indicates data was not available due to limited number of participants to calculate the data. | 0.10 (0) | 0.13 (59) | 0.16 (43) | 0.26 (56) | 0.54 (169)

15. Secondary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) Following Single and Repeat Dose Administration of GSK2816126
Description: Blood samples were collected from participants for pharmacokinetic analysis including Cmax following single (Day 1) and repeat dose (Day 15) administration of GSK2816126. Pharmacokinetic analysis of GSK2816126 in Part 1 was conducted by non-compartmental methods. NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: as for outcome 11
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 3 | 4 | 10 | 12 | 7
Microgram per milliliter
  Day 1; n=2,1,1,1,3,4,10,12,7 | 0.42 (52) | 1.10 (NA) — NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. | 1.40 (NA) — NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. | 4.00 (NA) — NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. | 7.31 (16) | 10.91 (10) | 13.04 (27) | 22.26 (35) | 23.83 (21)
  Day 15; n=1,1,1,1,3,4,9,11,4: number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 4 | 9 | 11 | 4
  Day 15; n=1,1,1,1,3,4,9,11,4 | 0.50 (NA) — NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. | 1.00 (NA) — NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. | 1.50 (NA) — NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. | 3.50 (NA) — NA indicates data was not available since geometric coefficient of variation could not be calculated for single participant. | 7.46 (13) | 11.62 (27) | 14.21 (27) | 21.62 (27) | 30.48 (14)

16. Secondary Outcome: Part 1: Time to Reach Cmax (Tmax) Following Single and Repeat Dose Administration of GSK2816126
Description: Blood samples were collected from participants for pharmacokinetic analysis including Tmax following single (Day 1) and repeat dose (Day 15) administration of GSK2816126. Tmax is the time to reach Cmax, determined directly from the concentration-time data. Pharmacokinetic analysis of GSK2816126 in Part 1 was conducted by non-compartmental methods. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: as for outcome 11
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 3 | 4 | 10 | 12 | 7
Hours
  Day 1; n=2,1,1,1,3,4,10,12,7 | 1.50 [1.0 to 2.0] | 1.00 [1.0 to 1.0] | 2.00 [2.0 to 2.0] | 1.90 [1.9 to 1.9] | 1.00 [0.5 to 1.9] | 2.05 [1.1 to 72.0] | 1.95 [1.0 to 2.9] | 2.00 [0.8 to 2.8] | 2.00 [0.5 to 3.3]
  Day 15; n=1,1,1,1,3,4,9,11,4: number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 4 | 9 | 11 | 4
  Day 15; n=1,1,1,1,3,4,9,11,4 | 2.70 [2.7 to 2.7] | 2.00 [2.0 to 2.0] | 1.00 [1.0 to 1.0] | 1.00 [1.0 to 1.0] | 2.00 [1.9 to 2.0] | 2.05 [2.0 to 2.1] | 1.90 [0.5 to 2.7] | 2.00 [1.0 to 3.0] | 2.25 [2.0 to 3.0]

17. Secondary Outcome: Part 1: Apparent Terminal Phase Elimination Rate Constant (Lambda z) Following Single and Repeat Dose Administration of GSK2816126
Description: Blood samples were collected from participants for pharmacokinetic analysis including lambda z following single (Day 1) and repeat dose (Day 15) administration of GSK2816126. Pharmacokinetic analysis of GSK2816126 in Part 1 was conducted by non-compartmental methods. Pharmacokinetic parameter derivation for some participants did not strictly conform to the prescribed acceptance criteria and hence data was not available for those participants. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: as for outcome 11
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours^-1
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 3 | 4 | 10 | 12 | 7
Hours^-1
  Day 1; n=2,0,0,1,3,1,10,10,7: number analyzed (Participants) | 2 | 0 | 0 | 1 | 3 | 1 | 10 | 10 | 7
  Day 1; n=2,0,0,1,3,1,10,10,7 | 0.15 [0.1 to 0.2] |  |  | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.1]
  Day 15; n=1,1,0,1,2,4,9,11,4: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2 | 4 | 9 | 11 | 4
  Day 15; n=1,1,0,1,2,4,9,11,4 | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] |  | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.1] | 0.00 [0.0 to 0.1] | 0.00 [0.0 to 0.0]

18. Secondary Outcome: Part 1: Apparent Terminal Phase Half-life (T1/2) Following Single and Repeat Dose Administration of GSK2816126
Description: Blood samples were collected from participants for pharmacokinetic analysis including T1/2 following single (Day 1) and repeat dose (Day 15) administration of GSK2816126. Pharmacokinetic analysis of GSK2816126 in Part 1 was conducted by non-compartmental methods. Pharmacokinetic parameter derivation for some participants did not strictly conform to the prescribed acceptance criteria and hence data was not available for those participants. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: as for outcome 11
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 3 | 4 | 10 | 12 | 7
Hours
  Day 1; n=2,0,0,1,3,1,10,10,7: number analyzed (Participants) | 2 | 0 | 0 | 1 | 3 | 1 | 10 | 10 | 7
  Day 1; n=2,0,0,1,3,1,10,10,7 | 8.90 [4.3 to 13.5] |  |  | 49.10 [49.1 to 49.1] | 27.20 [19.4 to 35.2] | 14.10 [14.1 to 14.1] | 32.55 [23.0 to 39.0] | 32.10 [25.6 to 48.8] | 21.80 [8.5 to 45.3]
  Day 15; n=1,1,0,1,2,4,9,11,4: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2 | 4 | 9 | 11 | 4
  Day 15; n=1,1,0,1,2,4,9,11,4 | 46.50 [46.5 to 46.5] | 36.80 [36.8 to 36.8] |  | 39.70 [39.7 to 39.7] | 27.40 [25.7 to 29.1] | 26.85 [23.0 to 33.8] | 30.00 [12.2 to 65.7] | 25.70 [8.2 to 38.3] | 30.20 [15.1 to 40.3]

19. Secondary Outcome: Part 1: Accumulation Ratio Following Administration of GSK2816126
Description: Accumulation ratio was determined from the ratio of AUC (0-tau) on Cycle 1 Day 15/AUC (0-tau) on Cycle 1 Day 1 by dose cohort. Only those participants with data available at the specified data points were analyzed. To assess accumulation ratio for a dose level based on ANOVA method, it was required that at least 2 participants had derived PK parameter AUC(0- tau) on both Cycle 1 Day 1 and Cycle 1 Day 15. For dose 100mg, 200mg and 400mg, only 1 participant received treatment. For dose 50mg, 2 participants received treatment but there was one participant whose AUC(0- tau) on Cycle 1 Day 15 could not be derived due to discontinuation of treatment before Day 15. Hence, accumulation ratio could not be calculated for these 4 arms. Accumulation ratio of GSK2816126 was estimated by calculating the ratio of geometric least squares (GLS) means of the AUC between Day 15 and Day 1 for all dose levels and corresponding 90 percent (%) confidence interval (CI) for each ratio.
Time Frame: as for outcome 11
Population: Pharmacokinetic Population. To assess accumulation ratio by ANOVA, it requires at least 2 participants to derive PK parameter AUC(0- tau) on both Cycle 1 Day 1 and Cycle 1 Day 15 which was not observed for dose 50mg, 100mg, 200mg and 400mg. Hence data could not be calculated for these 4 arms.
Measure: Number (90% Confidence Interval); unit: Ratio of AUC
Arm/Group | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 3 | 4 | 9 | 11 | 4
Ratio of AUC | 1.090 [0.827 to 1.435] | 0.625 [0.291 to 1.345] | 1.288 [1.173 to 1.415] | 1.224 [1.081 to 1.386] | 1.801 [0.819 to 3.959]

20. Secondary Outcome: Part 1: Time Invariance Ratio Following Administration of GSK2816126
Description: Ratio of AUC(0-tau) on Day15/Day1 AUC(0-inf) was calculated to assess time invariance. Only those participants with data available at specified data points were analyzed. To assess time invariance based on ANOVA method, it is required that at least 2 participants in a dose level had AUC(0-inf) on Cycle1 Day1 and AUC(0-tau) on Cycle1 Day15. For dose 100mg, 200mg and 400mg, only 1 participant received treatment. For 50mg, 2 participants received treatment but there was one participant whose AUC(0-tau) on Cycle1 Day15 could not be derived due to discontinuation of treatment before Day15, so time invariance could not be calculated. For 1200mg, 4 participants received treatment, however, AUC(0-inf) derivation on Cycle1 Day1 for 3 out of 4 participants did not strictly conform to the prescribed acceptance criteria. Time invariance ratio of GSK2816126 was estimated by calculating ratio of GLS means of AUC between Day15 and Day1 for all dose levels and corresponding 90% CI for each ratio.
Time Frame: as for outcome 11
Population: Pharmacokinetic Population. To assess time invariance by ANOVA, it requires at least 2 participants to have AUC(0-inf) and AUC(0-tau) on Cycle1 Day15 which was not observed for dose 50mg, 100mg, 200mg, 400mg. For 1200mg, AUC(0-inf) on Cycle1 Day1 for 3 participants did not meet acceptance criteria. Data could not be calculated for these 5 arms.
Measure: Number (90% Confidence Interval); unit: Ratio of AUC
Arm/Group | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 3 | 9 | 9 | 4
Ratio of AUC | 1.016 [0.814 to 1.269] | 1.157 [1.074 to 1.247] | 1.091 [0.937 to 1.269] | 1.606 [0.806 to 3.198]

21. Secondary Outcome: Part 1: Exposure Producing 50 Percent of the Maximum Effect (EC50) of GSK2816126 With Respect to Exposure Markers
Description: The pharmacokinetic/pharmacodynamic relationship between GSK2816126 exposure markers (dose, concentration, Cmax or AUC) was planned to be characterized by linear and/or non-linear mixed effect models. This analysis was planned to be based on Pharmacodynamic Population which consists of participants in the All Subjects population for whom a pharmacodynamics/biomarkers sample was obtained and analyzed. This analysis was planned but not performed as the pharmacodynamic response was not observed and therefore a relationship between pharmacokinetic and pharmacodynamic parameters could not be determined.
Time Frame: Up to 3.2 years
Population: Pharmacodynamic Population. Analysis was not performed as pharmacodynamic response was not observed.
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Part 1: Maximum Effect (Emax) of GSK2816126 With Respect to Exposure Markers
Description: The pharmacokinetic/pharmacodynamic relationship between GSK2816126 exposure markers (dose, concentration, Cmax or AUC) was characterized by linear and/or non-linear mixed effect models. This analysis was planned but not performed as the pharmacodynamic response was not observed and therefore a relationship between pharmacokinetic and pharmacodynamic parameters could not be determined.
Time Frame: Up to 3.2 years
Population: Pharmacodynamic Population. Analysis was not performed as pharmacodynamic response was not observed.
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Part 1: Number of Participants With Overall Change in Tri-methylated Histone H3 Lysine 27 (H3K27me3) Ratios Compared to Baseline
Description: The pre and post-treatment samples for tumor or surrogate tissue/body fluid (e.g. Peripheral blood mononuclear cell [PBMCs], blood, skin or hair) were collected for the analysis of H3K27me3. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Change from Baseline was defined as any visit value minus Baseline value.
Time Frame: Baseline and up to 3.2 years
Population: Pharmacodynamic Population
Measure: Number; unit: Participants
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 3 | 4 | 10 | 12 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Part 1: Percentage of Participants With Solid Tumors Achieving Best Overall Response Rate
Description: Overall response rate is defined as percentage of participants achieving complete response and partial response per RECIST version 1.1. Complete Response is the disappearance of all target/non-target lesions. Partial Response is at least a 30 percent decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters. The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence. The percentage of participants with solid tumors (including prostate) achieving best overall response rate have been presented. No participants with solid tumors were treated at doses below 800mg (i.e. 50mg, 100mg, 200mg, 400mg). Hence data could not be calculated for these 4 arms.
Time Frame: Up to 3.2 years
Population: All Subjects Population.Only those participants with data available at specific time point were analyzed. No participants with solid tumors were treated at doses below 800mg (i.e. 50mg, 100mg, 200mg, 400mg). Hence data could not be calculated for these 4 arms.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 1 | 2 | 5 | 8 | 5
Percentage of participants | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Part 1: Percentage of Participants With Lymphoma Achieving Best Overall Response Rate
Description: Overall response rate is defined as percentage of participants achieving complete response and partial response per RECIST version 1.1. Complete Response is the disappearance of all target/non-target lesions. Partial Response is at least a 30 percent decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters. The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence. The percentage of participants with lymphoma achieving best overall response rate have been presented.
Time Frame: Up to 3.2 years
Population: All Subjects Population
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 2 | 2 | 5 | 4 | 2
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 0 | 0

26. Secondary Outcome: Part 1: Concentration of GSK2816126 and Its Metabolites in Blood
Description: Blood samples were planned to be collected from participants in the pharmacokinetic/pharmacodynamic expansion cohort for analysis of GSK2816126 and its metabolites. Samples were not collected due to early termination of the study; therefore, no analysis could be performed.
Time Frame: as for outcome 11
Population: Pharmacokinetic Population. Samples were not collected due to early study termination.
Groups:
- Part 1: Participants With GCB-DLBCL: At maximum tolerated or recommended phase II dose, participants with GCB-DLBCL were enrolled in Part 1 expansion cohorts and received GSK2816126 twice-weekly, as intravenous solution.
- Part 1: Participants With Solid Tumors: At maximum tolerated or recommended phase II dose, participants with solid tumors were enrolled in Part 1 expansion cohorts and received GSK2816126 twice-weekly, as intravenous solution.
Arm/Group | Part 1: Participants With GCB-DLBCL | Part 1: Participants With Solid Tumors
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Part 1: Concentration of GSK2816126 and Its Metabolites in Bile
Description: Bile samples were planned to be collected from participants in the pharmacokinetic/pharmacodynamic expansion cohort for analysis of GSK2816126 and its metabolites via the Entero-Test. Samples were not collected due to early termination of the study; therefore, no analysis could be performed.
Time Frame: Day 15
Population: Pharmacokinetic Population. Samples were not collected due to early study termination.
Arm/Group | Part 1: Participants With GCB-DLBCL | Part 1: Participants With Solid Tumors
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Part 1: Concentration of GSK2816126 and Its Metabolites in Urine
Description: Urine samples were planned to be collected from participants in the pharmacokinetic/pharmacodynamic expansion cohort for analysis of GSK2816126 and its metabolites. Samples were not collected due to early termination of the study; therefore, no analysis could be performed.
Time Frame: Pre-dose and 0 to 24 hours post-dose on Day 1; 0 to 8 hours post-dose on Day 15
Population: Pharmacokinetic Population. Samples were not collected due to early study termination.
Arm/Group | Part 1: Participants With GCB-DLBCL | Part 1: Participants With Solid Tumors
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Part 1:Concentration of GSK2816126 in Urine After Dosing at Steady State
Description: The amount of GSK2816126 excreted in urine after dosing at steady state was determined. The concentration of GSK2816126 in urine was planned to be measured with an investigational bio-analytical method and extrapolated to total amount excreted in urine over time using urine volume. Samples were not collected due to early termination of the study; therefore, no analysis could be performed.
Time Frame: Pre-dose and 0 to 24 hours post-dose on Day 1; 0 to 8 hours post-dose on Day 15
Population: Pharmacokinetic Population Samples were not collected due to early study termination.
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

30. Secondary Outcome: Part 2: Number of Participants With SAEs and Non-SAEs
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/ incapacity, is a congenital anomaly/ birth defect, other situations and is associated with liver injury or impaired liver function. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 3.2 years
Population: All Subjects Population. Data was not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

31. Secondary Outcome: Part 2: Number of Participants With DLTs
Description: An event was considered a DLT if it occurred within first 4 weeks (28 days) of treatment, and met the criteria's for hematologic , non-hematologic, infusion reactions and other toxicities, unless it can be clearly established that the event is unrelated to treatment. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 4 weeks
Population: All Subjects Population. Data was not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

32. Secondary Outcome: Part 2: Number of Participants Withdrawn Due to AEs
Description: A participant was considered to have completed the study if they have completed their end of study visit or if the participant died or was still in follow-up at the time the study was closed or terminated. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 3.2 years
Population: All Subjects Population. Data was not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

33. Secondary Outcome: Part 2: Number of Participants With Dose Interruptions
Description: The number of participants who had any dose interruptions were planned to be analyzed. However, this analysis was not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 3.2 years
Population: All Subjects Population. Data was not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

34. Secondary Outcome: Part 2: Number of Participants With Dose Reductions
Description: The number of participants who had any dose reduction or delay were planned to be analyzed. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 3.2 years
Population: All Subjects Population. Data was not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

35. Secondary Outcome: Part 2: Number of Participants With Worst Case Change From Baseline in Clinical Chemistry Parameters
Description: Blood samples were planned to be collected for evaluation of clinical chemistry parameters including direct bilirubin, chloride, LDH, total protein, urea/BUN and uric acid. Baseline value was defined as the most recent, non-missing value from a local laboratory prior to the first dose of study treatment. Change from Baseline was defined as any visit value minus Baseline value. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Baseline and up to 3.2 years
Population: All Subjects Population. Data was not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

36. Secondary Outcome: Part 2: Number of Participants With Worst Case Changes From Baseline in Hematology Parameters
Description: Blood samples were planned to be collected for the analysis of hematology parameters including basophils, eosinophils, hematocrit, MCHC, MCH, MCV, monocytes, seg neutrophils, RBC count and reticulocytes. Baseline value was defined as the most recent, non-missing value from a local laboratory prior to the first dose of study treatment. Change from Baseline was defined as any visit value minus Baseline value. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Baseline and up to 3.2 years
Population: All Subjects Population. Data was not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

37. Secondary Outcome: Part 2: Number of Participants With Abnormal Values for Vital Signs
Description: Vital sign measurements includes SBP, DBP, body temperature and heart rate. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 3.2 years
Population: All Subjects Population. Data was not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

38. Secondary Outcome: Part 2: Number of Participants With Abnormal Findings for ECG Parameters
Description: Single measurements of 12-lead ECGs were planned to be obtained a semi-recumbent or semi-supine position after at least a 5 minutes rest using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT and QTc intervals. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 3.2 years
Population: All Subjects Population. Data was not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

39. Secondary Outcome: Part 2: Clearance Following Administration of GSK2816126
Description: Blood samples were planned to be collected at Pre-dose, single draw between 0.5 and 1.9 hours from start of infusion, single draw between 3-6 hours following end of infusion on Day 1 and Day 11; Pre-dose on Day 4; Day 8, Day 11; Pre-dose on Day 15 for Cycle 1 and Cycles 2, 4, 6 and 12 pre-dose and within 5 minutes prior to end of infusion on Day 4 for population pharmacokinetic analysis of GSK2816126 including clearance. Each cycle was of 28 days. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 3.2 years
Population: Pharmacokinetic Population. Data was not collected in Part2 as no participant was enrolled in Part2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

40. Secondary Outcome: Part 2: Volume of Distribution Following Administration of GSK2816126
Description: Blood samples were planned to be collected on Pre-dose, single draw between 0.5 and 1.9 hours from start of infusion, single draw between 3-6 hours following end of infusion on Day 1 and Day 11; Pre-dose on Day 4; Day 8,Day 11; Pre-dose on Day 15 for Cycle 1 and Cycle 2, 4, 6 and 12 pre-dose and within 5 minutes prior to end of infusion on Day 4 for population pharmacokinetic analysis of GSK2816126 including clearance. Each cycle was of 28 days. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 3.2 years
Population: Pharmacokinetic Population. Data was not collected in Part2 as no participant was enrolled in Part2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

41. Secondary Outcome: Part 2:EC50 of GSK2816126 With Respect to Exposure Markers
Description: The pharmacokinetic/pharmacodynamic relationship between GSK2816126 exposure markers (dose, concentration, Cmax or AUC) was planned to be characterized by linear and/or non-linear mixed effect models. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 3.2 years
Population: Pharmacodynamic Population. Data was not collected in Part2 as no participant was enrolled in Part2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

42. Secondary Outcome: Part 2:Emax of GSK2816126 With Respect to Exposure Markers
Description: as for outcome 41
Time Frame: Up to 3.2 years
Population: Pharmacodynamic Population. Data was not collected in Part2 as no participant was enrolled in Part2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

43. Secondary Outcome: Part 2: Number of Participants With Change in H3K27me3 Ratios Compared to Baseline
Description: The pre and post-treatment samples for tumor or surrogate tissue/body fluid (e.g. PBMCs, blood, skin or hair) were planned to be collected for the analysis of H3K27me3. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Change from Baseline was defined as any visit value minus Baseline value. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Baseline and up to 3.2 years
Population: Pharmacodynamic Population. Data was not collected in Part2 as no participant was enrolled in Part2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

44. Secondary Outcome: Part 2: Concentration of GSK2816126 and Its Metabolites in Blood
Description: Blood samples were planned to be collected from participants in the pharmacokinetic/pharmacodynamic expansion cohort for analysis of GSK2816126 and its metabolites. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Pre-dose, single draw between 0.5 and 1.9 hours from start of infusion, single draw between 3-6 hours following end of infusion on Day 1; Pre-dose on Day 15 for Cycle 1 and Cycles 2, 4, 6 and 12 (Each cycle was of 28 days)
Population: Pharmacokinetic Population. Data was not collected in Part2 as no participant was enrolled in Part2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

45. Secondary Outcome: Part 2: Concentration of GSK2816126 and Its Metabolites in Bile
Description: Bile samples were planned to be collected from participants in the pharmacokinetic/pharmacodynamic expansion cohort for analysis of GSK2816126 and its metabolites via the Entero-Test. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Day 15
Population: Pharmacokinetic Population. Data was not collected in Part2 as no participant was enrolled in Part2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

46. Secondary Outcome: Part 2: Concentration of GSK2816126 and Its Metabolites in Urine
Description: Urine samples were planned to be collected from participants in the pharmacokinetic/pharmacodynamic expansion cohort for analysis of GSK2816126 and its metabolites. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Pre-dose and 0 to 24 hours post-dose on Day 1; 0 to 8 hours post-dose on Day 15
Population: Pharmacokinetic Population. Data was not collected in Part2 as no participant was enrolled in Part2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

47. Secondary Outcome: Part 2:Concentration of GSK2816126 in Urine After Dosing at Steady State
Description: The amount of GSK2816126 excreted in urine after dosing at steady state was planned to be determined. The concentration of GSK2816126 in urine was planned to be measured with an investigational bio-analytical method and extrapolated to total amount excreted in urine over time using urine volume. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Pre-dose and 0 to 24 hours post-dose on Day 1; 0 to 8 hours post-dose on Day 15
Population: Pharmacokinetic Population. Data was not collected in Part2 as no participant was enrolled in Part2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

48. Secondary Outcome: Part 2: Change in 4-beta-hydroxy Cholesterol to Cholesterol Ratio From Baseline Following Repeat Dosing of GSK2816126
Description: Plasma analysis for 4-beta-hydroxycholesterol and cholesterol was planned to be conducted. Baseline value was defined as the most recent, non-missing value from a local laboratory prior to the first dose of study treatment. Change from Baseline was defined as any visit value minus Baseline value. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Baseline and up to 21 days
Population: Pharmacodynamic Population. Data was not collected in Part2 as no participant was enrolled in Part2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

49. Secondary Outcome: Part 2: Duration of Response
Description: Duration of response for participants is defined as the time from the first documented evidence of a PR or CR until the first documented sign of disease progression or death due to any cause. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 3.2 years
Population: All Subjects Population. Data was not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

50. Secondary Outcome: Part 2: Number of Participants With Progression Free Survival
Description: PFS is defined as the interval between the first dose of study medication and the earliest date of disease progression or death due to any cause. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 3.2 years
Population: All Subjects Population. Data was not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2: All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (Non-SAEs) were collected in Part 1 from the start of the study treatment up to 3.2 years.
Description: SAEs and Non-SAEs were collected in Part A from All Subjects Population which included all participants who receive at least one dose of study treatment. Data were not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 1:GSK2816126 50 mg Twice-weekly | Part 1:GSK2816126 100 mg Twice-weekly | Part 1:GSK2816126 200 mg Twice-weekly | Part 1:GSK2816126 400 mg Twice-weekly | Part 1:GSK2816126 800 mg Twice-weekly | Part 1:GSK2816126 1200 mg Twice-weekly | Part 1:GSK2816126 1800 mg Twice-weekly | Part 1:GSK2816126 2400 mg Twice-weekly | Part 1:GSK2816126 3000 mg Twice-weekly | Part 2: All Participants
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/1 | 0/1 | 0/1 | 0/3 | 1/4 | 2/10 | 0/12 | 1/7 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/1 | 0/1 | 0/1 | 1/3 | 2/4 | 1/10 | 5/12 | 3/7 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 1/1 | 1/1 | 3/3 | 4/4 | 10/10 | 12/12 | 7/7 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1:GSK2816126 50 mg Twice-weekly (N=2) | Part 1:GSK2816126 100 mg Twice-weekly (N=1) | Part 1:GSK2816126 200 mg Twice-weekly (N=1) | Part 1:GSK2816126 400 mg Twice-weekly (N=1) | Part 1:GSK2816126 800 mg Twice-weekly (N=3) | Part 1:GSK2816126 1200 mg Twice-weekly (N=4) | Part 1:GSK2816126 1800 mg Twice-weekly (N=10) | Part 1:GSK2816126 2400 mg Twice-weekly (N=12) | Part 1:GSK2816126 3000 mg Twice-weekly (N=7) | Part 2: All Participants (N=0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Campylobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1:GSK2816126 50 mg Twice-weekly (N=2) | Part 1:GSK2816126 100 mg Twice-weekly (N=1) | Part 1:GSK2816126 200 mg Twice-weekly (N=1) | Part 1:GSK2816126 400 mg Twice-weekly (N=1) | Part 1:GSK2816126 800 mg Twice-weekly (N=3) | Part 1:GSK2816126 1200 mg Twice-weekly (N=4) | Part 1:GSK2816126 1800 mg Twice-weekly (N=10) | Part 1:GSK2816126 2400 mg Twice-weekly (N=12) | Part 1:GSK2816126 3000 mg Twice-weekly (N=7) | Part 2: All Participants (N=0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 6 (6) | 7 (7) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 3 (6) | 9 (10) | 3 (6) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 6 (6) | 5 (5) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 6 (6) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 2 (4) | 2 (2) | 3 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (11) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (3) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal paraesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood uric acid decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling of body temperature change (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated prior to the completion of Part 1 due to an unfavorable benefit risk profile. Part 2 was never initiated and no participants were enrolled. Participants time on treatment was for a maximum 210 days and a median of 56 days.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT02082977/SAP_000.pdf
  • Study Protocol (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT02082977/Prot_001.pdf